CLINICAL TRIAL: NCT01475110
Title: Observational Study in Adult Patients With Imatinib-resistant or Intolerant Chronic Myeloid Leukemia (CML) Treated With Nilotinib: Follow-up of the Italian Patients. GIMEMA Study CML0609
Brief Title: Observational Study in Adults With Imatinib-resistant/Intolerant Chronic Myeloid Leukemia Treated With Nilotinib
Acronym: CML0609
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: CML0609
Record Dates: First submitted 2011-11-11; First posted 2011-11-21 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Chronic Myeloid Leukaemia
Keywords: Imatinib; Chronic Myeloid Leukaemia; Nilotinib; Adult patients; Imatinib resistant
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study cohort group: Adult patients with Imatinib resistant (failure + suboptimal) or intolerant chronic myeloid leukaemia in all phases, who started treatment with Nilotinib between January 2005 and December 2012 in Italy.
  Adult pts treated with Nilotinib as second line therapy after Dasatinib.
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Observation of Imatinib resistant patients treated with Nilotinib.

SUMMARY:
The GIMEMA CML Working Party promotes an observational (retrospective and perspective) study of Imatinib-resistant or intolerant CML patients treated with Nilotinib in Italy. Enrollment will include all patients who started Nilotinib between January 2005 and December 2012. Patients will be followed for 4 years since treatment start. After this time, survival data, disease status and treatment will be recorded at 6-months-interval. This study will help the definition of guidelines for a proper management of Nilotinib in any-phase CML patients.

DETAILED DESCRIPTION:
Follow-up is required until the end of treatment for the purposes of the study for all patients by standard hematologic, cytogenetic and molecular criteria. This study will not contemplate any additional expense beyond what is expected for a regular follow-up, according to the international guidelines for CML.

Sample Size: target accrual was not defined, all eligible patients observed between January 2005 and December 2012 will be included.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Imatinib resistant (failure + suboptimal) or intolerant chronic myeloid leukaemia in all phases, who started treatment with Nilotinib between January 2005 and December 2012 in Italy.
* Adult pts treated with Nilotinib as second line therapy after Dasatinib.

Exclusion Criteria:

* Patients less than 18 year old.
* Use of Nilotinib as first line treatment.
* Patients treated with Nilotinib before 2005.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The GIMEMA CML Working Party promotes an observational (retrospective and perspective) study of Imatinib-resistant or intolerant CML patients treated with Nilotinib in Italy. Enrollement will include all patients who started Nilotinib between January 2005 and December 2012.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-09-13 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2016-11-24 (Actual)

PRIMARY OUTCOMES:
Overall Survival | At one year from study entry

SECONDARY OUTCOMES:
Rate of complete haematologic remission t | At one year from study entry
  Rate of complete haematologic remission with Nilotinib treatment and the duration of the responses.
Nilotinib safety profile with time (grade 3-4 AE and of SAE) and causes of death | At one year from study entry
Event Free Survival (EFS) | At one year from study entry
Progression Free Survival (PFS) | At one year from study entry
Rate of point mutations before or after Nilotinib treatment | At one year from study entry
Rate of major cytogenetic response | At one year from study entry
  Rate of major cytogenetic response with Nilotinib treatment and the duration of the responses.
Rate of compete cytogenetic response | At one year from study entry
  Rate of complete cytogenetic response with Nilotinib treatment and the duration of the responses.
Rate of major molecular remission | At one year from study entry
  Rate of major molecular remission with Nilotinib treatment and the duration of the responses.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe SAGLIO, Pr., Principal Investigator — Divisione di Medicina Interna-Ematologia, Ospedale San Luigi Gonzaga, Regione Gonzole 10, 10043 Orbassano
Locations (33):
- Italy (33):
  - Centro Oncologico Basilicata, Rionero in Vulture, Potenza
  - Ospedale, Alessandria
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - S.G. Moscati Hospital, Avellino
  - Ospedale, Bari
  - Ospedale, Bologna
  - Azienda Spedali Civili, Brescia
  - Ospedale Ferrarotto, Catania
  - Sez.Ematologia e Dip. scienze Biomediche Arcispedale S. Anna, Ferrara
  - Policlinico di Careggi, Università delgi studi di Firenze, Florence
  - Clinica Ematologica - Università degli Studi, Genova
  - Università degli Studi, Genova
  - Università di Genova, Genova
  - ASL Le1 P.O. Vito Fazzi - U.O. di Ematologia, Lecce
  - A.O. Universitaria Policlinico Martina di Messina, Messina
  - U.O. Ematologia e Trapianto di Midollo - Ist. Scientifico Ospedale San Raffaele, Milan
  - Federico II, Napoli
  - Divisione di Medicina Interna-Ematologia, Ospedale San Luigi Gonzaga, Regione Gonzole 10, Orbassano
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale Cervello, Palermo
  - Azienda Ospedaliera Universitaria - Policlinico Paolo Giaccone, Palermo
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Ospedale, Reggio Calabria
  - Ospedale, Rimini
  - U.O. di Ematologia - Centro Oncologico Basilicata, Rionero in Vulture
  - Ematologia - Sapienza Università di Roma, Roma
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O. Ematologia, Azienda Ospedaliera Universitaria Senese, Siena
  - Ospedale, Taranto
  - SCDO Ematologia 2 AOU S. Giovanni Battista, Torino
  - Policlinico Universitario - Clinica Ematologia, Udine
  - Policlinico G. B. Rossi - Borgo Roma, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation Website — http://www.gimema.it